CLINICAL TRIAL: NCT02861495
Title: Humeral Compression/Distraction (CD) Device Used for Fixation of Humeral Fractures
Brief Title: Humeral Compression/Distraction Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to low enrollment.
Sponsor: Florida Orthopaedic Institute (Network)
Collaborators: NuVasive (Industry); St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001
Record Dates: First submitted 2016-08-03; First posted 2016-08-10 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Humeral Fractures
Keywords: upper extremity fracture
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- humeral nail (Experimental): Surgical fixation with a humeral compression/distraction nail.
  Interventions: Device: Humeral Compression/Distraction (CD) Nail

INTERVENTIONS:
Device: Humeral Compression/Distraction (CD) Nail — Surgical fixation of humeral shaft fractures with Humeral Compression/Distraction (CD) Nail implant

SUMMARY:
The proposed study of humeral shaft fractures in adults will examine outcomes in patients treated with the Humeral Trauma Nail System to treat displaced humeral shaft fractures (displaced OTA code 12A, B, or C), nonunions, or malunions. The device to be studied uses an internal gear system controlled wirelessly by rare earth magnets, which typically offers distraction for lengthening. In the humerus however, during the treatment of acute fractures, this percutaneously inserted nail can also offer compression during the healing process, thereby negating the effect of gravity, which may in turn lead to a faster and more consistent rate of union. Furthermore, in cases of slower healing the dynamic properties of the nail may employ an "accordion technique" (alternating compression-distraction, a feature unique to this implant.

DETAILED DESCRIPTION:
The primary end point will be the union rate without secondary procedures. The hypothesis is that with the compression and distraction that this device makes possible, the investigators can achieve a higher union rate than with other forms of treatment, using a percutaneous approach, with a decreased complication rate, and can dynamically modulate the healing response when needed. The primary safety endpoint is the occurrence of adverse events from the time of treatment.

During the healing process an external remote controller (ERC) will be used to continually compress or distract the fracture as needed. The surgeon will monitor healing and decide, clinically based on sequential radiographs during subsequent office visits, whether the fracture needs additional compression or distraction, an accordion technique, or no additional external manipulation via the ERC. Participants will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult skeletally mature patients 18 years or older, treated by the Orthopaedic Trauma Service at Tampa General Hospital, and the Trauma Service at St. Louis University Hospital

  * Open or closed displaced humeral shaft fractures (displaced OTA code 12A, B, or C), nonunions or malunions
  * amenable to treatment with an intramedullary nail

Exclusion Criteria:

* Intra-articular extension of the fracture, prohibiting treatment with an intramedullary nail;
* Pathologic fracture
* Retained hardware
* Patients with pacemakers
* Age under 18 years.
* Patients who are prisoners or likely to become prisoners
* Homeless, or those likely to have difficulty making follow-up appointments
* Pregnancy
* Ipsilateral nerve or vascular injuries
* Immunocompromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Union rate | 3 months post operatively
  Union rate for compression/distraction nail will be compared to retrospective cohort of surgical fixation with humeral plates.

SECONDARY OUTCOMES:
Complication rate | 12 months
  Complication rate for compression/distraction nail will be compared to retrospective cohort of surgical fixation with humeral plates.
Adverse Events | 12 months
  Adverse event rate for compression/distraction nail will be compared to retrospective cohort of surgical fixation with humeral plates.

CONTACTS AND LOCATIONS:
Overall Officials: Roy W Sanders, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data at this time.